CLINICAL TRIAL: NCT05476549
Title: Effects of Lemon Verbena Extract Supplementation on Behaviour Mood and Cognitive Function in Sub-ADHD Children
Brief Title: Effects of Lemon Verbena Extract Supplementation in Sub-ADHD Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Finzelberg GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 48CD1
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Behavior, Child; Cognitive Change
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lemon verbena (Experimental)
  Interventions: Dietary Supplement: Lemon verbena
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lemon verbena — Lemon verbena supplement administered at an estimated daily dose of 15mg/kg
  Arms: Lemon verbena
Dietary Supplement: Placebo — Placebo supplement containing carrier material only
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the effects of 15 mg/kg lemon verbena, in comparison to placebo, on the attention deficit hyperactivity disorder (ADHD) type behaviour and cognitive function of children who do not have a diagnosis of ADHD, but who exhibit high scores (highest tertile) on ADHD behaviour parameters. Multiple aspects of mood will also be assessed.

The proposed randomised, double-blind, placebo-controlled, parallel groups design methodology will assess the psychological effects of 15 mg/kg lemon verbena extract and a matched placebo prior to and after 4 and 8 weeks of supplementation. The trial will utilise the COMPASS cognitive assessment system (Northumbria University) and a range of mood measures during laboratory testing visits.

Parents and children will also take part in a concomitant smartphone study, comprising the collection of the parent's assessment of the child's behaviour/cognitive function and the child's self-report of the same, plus their mood. These assessments will take place on Days -1, 14, 28, 42 and 56.

ELIGIBILITY:
Inclusion Criteria:

* Are in good health as reported by themselves and their parent/guardian
* Are aged 8 to 17 years at the time of giving assent and parents giving consent
* Have a sex and age-related BMI less than the 98th centile according to the local NHS guidelines
* Are rated by their parents as having a high score (T score of ≥60) on both the Connors 3 subscales of Inattention and Hyperactivity/Impulsivity.
* Have no current diagnosis of ADHD
* Have no relevant food intolerances/ sensitivities/ allergies
* Are not currently using any illicit, herbal or recreational drugs including alcohol and nicotine products
* Are not currently taking prescription medications
* Have not taken dietary supplements e.g. Vitamins, omega 3 fish oils etc. in the last 4 weeks
* Do not have a diagnosed neurological condition, or learning/behavioural or neurodevelopmental differences (e.g. dyslexia, autism)
* Do not suffer from visual (including colour blindness) impairment that cannot be corrected with glasses or lenses (that may impact task performance in the opinion of the PI).
* Do not have any pre-existing diagnosed medical condition/illness which will impact taking part in the study
* Consume less than 250 mg/day of caffeine.
* Can complete all of the study assessments at the training visit
* Are not currently participating in other clinical or nutrition intervention studies, or have in the past 4 weeks
* Are compliant with regards to treatment consumption
* Have not taken antibiotics within the past 4 weeks
* Do not have any health condition that would prevent fulfilment of the study requirements (this includes non-diagnosed conditions for which no medication may be taken)

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2023-08-27 (Actual); Study Completion 2023-08-27 (Actual)

PRIMARY OUTCOMES:
Change in Conners 3 score from baseline to 8 weeks, parent rating | Baseline to 8 weeks
Change in Conners 3 score from baseline to 8 weeks, child rating | Baseline to 8 weeks
Change in total mood disturbance from baseline to 8 weeks | Baseline to 8 weeks
  Profile of mood states questionnaire
Change in depression-dejection from baseline to 8 weeks | Baseline to 8 weeks
  Profile of mood states questionnaire
Change in tension-anxiety from baseline to 8 weeks | Baseline to 8 weeks
  Profile of mood states questionnaire
Change in anger-hostility from baseline to 8 weeks | Baseline to 8 weeks
  Profile of mood states questionnaire
Change in confusion-bewilderment from baseline to 8 weeks | Baseline to 8 weeks
  Profile of mood states questionnaire
Change in vigour-activity from baseline to 8 weeks | Baseline to 8 weeks
  Profile of mood states questionnaire
Change in fatigue-inertia from baseline to 8 weeks | Baseline to 8 weeks
  Profile of mood states questionnaire
Change in systolic blood pressure from baseline to 8 weeks | Baseline to 8 weeks
  Systolic blood pressure (mmHg)
Change in diastolic blood pressure from baseline to 8 weeks | Baseline to 8 weeks
  Diastolic blood pressure (mmHg)
Change in body temperature from baseline to 8 weeks | Baseline to 8 weeks
  Degrees Celsius
Change in RMSSD during the performance of cognitive tasks from baseline to 8 weeks | Baseline to 8 weeks
  Root mean square of successive differences between normal heartbeats (RMSSD)
Change in heart rate during the performance of cognitive tasks from baseline to 8 weeks | Baseline to 8 weeks
  Beats per minute
Change in heart rate variability index during the performance of cognitive tasks from baseline to 8 weeks | Baseline to 8 weeks
  Heart rate variability index
Change in pNN50 during the performance of cognitive tasks from baseline to 8 weeks | Baseline to 8 weeks
  pNN50 is the mean number of times per hour in which the change in consecutive normal sinus (NN) intervals exceeds 50 milliseconds.
Change in stress index during the performance of cognitive tasks from baseline to 8 weeks | Baseline to 8 weeks
  The stress index is a measure of the ratio between the parasympathetic and sympathetic tone. intervals exceeds 50 milliseconds.
Change in subjective anxiety from baseline to 8 weeks | Baseline to 8 weeks
  State-trait anxiety inventory (STAI) total score
Change in subjective perceived stress from baseline to 8 weeks | Baseline to 8 weeks
  Perceived stress scale (PSS) total score
Change in subjective mood from baseline to 8 weeks, alertness | Baseline to 8 weeks
  Visual analogue scale composite score
Change in subjective mood from baseline to 8 weeks, stress | Baseline to 8 weeks
  Visual analogue scale composite score
Change in subjective mood from baseline to 8 weeks, tranquility | Baseline to 8 weeks
  Visual analogue scale composite score
Change in speed of performance from baseline to 8 weeks | Baseline to 8 weeks
  Cognitive task composite score, milliseconds
Change in accuracy of performance from baseline to 8 weeks | Baseline to 8 weeks
  Cognitive task composite score, %
Change in accuracy of performance on arrow flankers task from baseline to 8 weeks | Baseline to 8 weeks
  Cognitive task score, %
Change in accuracy of performance on numeric working memory task from baseline to 8 weeks | Baseline to 8 weeks
  Cognitive task score, %
Change in accuracy of performance on Stroop task from baseline to 8 weeks | Baseline to 8 weeks
  Cognitive task score, %
Change in accuracy of performance on Corsi blocks task from baseline to 8 weeks | Baseline to 8 weeks
  Cognitive task score, %
Change in accuracy of performance on rapid visual information processing task from baseline to 8 weeks | Baseline to 8 weeks
  Cognitive task score, %
Change in accuracy of performance on peg and ball task from baseline to 8 weeks | Baseline to 8 weeks
  Cognitive task score, number of errors
Change in reaction time of performance on arrow flankers task from baseline to 8 weeks | Baseline to 8 weeks
  Cognitive task score, reaction time in milliseconds
Change in reaction time of performance on numeric working memory task from baseline to 8 weeks | Baseline to 8 weeks
  Cognitive task score, reaction time in milliseconds
Change in reaction time of performance on Stroop task from baseline to 8 weeks | Baseline to 8 weeks
  Cognitive task score, reaction time in milliseconds
Change in reaction time of performance on rapid visual information processing task from baseline to 8 weeks | Baseline to 8 weeks
  Cognitive task score, reaction time in milliseconds
Change in false alarms on rapid visual information processing task from baseline to 8 weeks | Baseline to 8 weeks
  Cognitive task score, number of false alarms
Change in completion time of peg and ball task from baseline to 8 weeks | Baseline to 8 weeks
  Cognitive task score, time in milliseconds
Change in thinking time of peg and ball task from baseline to 8 weeks | Baseline to 8 weeks
  Cognitive task score, time in milliseconds

CONTACTS AND LOCATIONS:
Overall Officials: Philippa Jackson, PhD, Principal Investigator — Northumbria University
Locations (1):
- Brain, Performance, Nutrition Research Centre, Northumbria University, Newcastle upon Tyne, Tyne & Wear, United Kingdom